CLINICAL TRIAL: NCT00655889
Title: Safety and Efficacy Study of Isolagen TherapyTM in Treatment of Interdental Papillary Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-G-003
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Interdental Papillary Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental)
  Interventions: Biological: Autologous Human Fibroblasts (azficel-T)

INTERVENTIONS:
Biological: Autologous Human Fibroblasts (azficel-T) — 1. Collection of biopsy from palate
  2. Papillary priming procedure
  3. Seven injection treatments to target sites
  4. Performance of study assessments (investigator and subject)
  Other Names: LAVIV

SUMMARY:
The purpose of this study is to evaluate the safety profile and the treatment effect of Isolagen TherapyTM in subjects with maxillary lesions who were treated in a previous study (IT-G-002, no NCT identification number)

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18-70 years of age
* Subject was treated in IT-G-002 (no NCT identification number)
* Subject has maxillary interproximal recession defects
* Natural teeth must be present on both sides of each area to be treated
* Negative pregnancy test and use of acceptable birth control (females of childbearing age)

Exclusion Criteria:

* Subjects who participated in other clinical trials within 30 days prior to enrollment
* Interproximal spaces including root grooves or furcations must not be involved
* Subjects with poor oral hygiene
* Subjects with a systemic condition, which would preclude periodontal treatment
* Subjects with acute infectious lesions in the treatment areas
* Subjects with open interproximal contact at study sites
* Subjects who must receive prophylactic antibiotics before dental procedures
* Subjects on chronic antibiotic or steroidal therapy
* Subjects with interproximal probing depths > 3 mm around study lesions
* Subjects who smoke
* Subjects taking medications associated with the development of drug induced gingival hyperplasia
* Subjects with radiographic evidence of pathology
* Subjects with tooth mobility exceeding a score of 1
* Subjects with parafunctional habits and not wearing bite guard
* Subjects with interproximal spaces associated with teeth without an adequate zone of keratinized tissue
* Subjects where the etiology of the interproximal papillary recession has not been controlled
* Subjects who have received a crown or pontic on one or both teeth involved in the interproximal space to be treated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Perio-Health Professionals, Inc., Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between July 17, 2006 to September 11, 2006.
Groups:
- Autologous Fibroblasts: Patients received autologous fibroblasts to maxillary interdental papillary recessions that were treated with fibroblasts or placebo in a previous study.
Period: Overall Study
Arm/Group | Autologous Fibroblasts
Started | 13
Completed | 11
Not Completed | 2
Not completed — Inadequate cell growth | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders Based on the Average Investigator Evaluation of Change From Baseline for All Treated Areas on the Global Ordinal Rating Scale (GORS)
Description: A patient was considered a responder in this outcome measure if the average Investigator's GORS score for all treatment areas was greater than 0. On the GORS, a score of -2 (much worsening from baseline) was the worst and +2 (great improvement from baseline) was the best.
Time Frame: Baseline (prior to first study treatment) compared to six months after first treatment
Population: Subjects who received at least one treatment during the study were included in the Intent to Treat population
Measure: Number; unit: participants
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 12
participants | 10

2. Primary Outcome: Number of Responders Based on the Average Patient Evaluation of Change From Baseline for All Treated Areas on the Global Ordinal Rating Scale (GORS)
Description: A patient was considered a responder in this outcome measure if the average patient's GORS score for all treatment areas was greater than 0. On the GORS, a score of -2 (much worsening from baseline) was the worst and +2 (great improvement from baseline) was the best.
Time Frame: Baseline (prior to first study treatment) compared to six months after first treatment
Population: Subjects who received at least one treatment during the study were included in the Intent to Treat population
Measure: Number; unit: participants
Arm/Group | Autologous Fibroblasts
Number analyzed (Participants) | 12
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for one year after first study treatment
Groups:
- Autologous Fibroblasts: Patients received autologous fibroblasts to maxillary interdental papillary recessions that were treated with fibroblasts or placebo in a previous study (IT-G-002, no NCT identification number).
Arm/Group | Autologous Fibroblasts
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblasts (N=13)
Appendicitis (Gastrointestinal disorders) | 1 (1) — Patient experienced an event of appendicitis. The event was considered unrelated to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblasts (N=13)
Accidental Injury (General disorders) | 1 (1)
Herpes Simplex (Skin and subcutaneous tissue disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Periodontal Abscess (Gastrointestinal disorders) | 1 (1)
Flu Syndrome (General disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a small, open-label study without a placebo control, and was not powered to provide statistically significant demonstrations of product efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications or presentations by the Investigator or his associates, were required to be submitted to the sponsor for review and approval prior to publication or presentation in any form.